CLINICAL TRIAL: NCT04808466
Title: Comparative Study on the Efficacy of Lobaplatin and Paclitaxel in the Treatment of Advanced Gastric Cancer Patients With D2 Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Comparative Study of Lobaplatin and Paclitaxel in Advanced Gastric Cancer Patients With D2 Surgery Combined With Hyperthermic Intraperitoneal Chemotherapy
Acronym: WUHIPEC01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHCT-IEC-SOP-016-21-01
Record Dates: First submitted 2021-02-17; First posted 2021-03-22 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer; Chemotherapy Effect; Surgery; Metastasis; Survival
Keywords: advanced gastric cancer; hyperthermic intraperitoneal chemotherapy; lobaplatin; paclitaxel; prognosis
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; lobaplatin

STUDY DESIGN:
Intervention Model Description: We divide patients into 3 groups randomly. Test group 1: D2 Surgery + HIPEC (paclitaxel) + SOX/XELOX regimen Test group 2: D2 Surgery + HIPEC (lobaplatin) + SOX/XELOX regimen Control group: D2 Surgery + HIPEC (no drug) + SOX/XELOX regimen
Who Masked: Participant
Masking Description: the choice of HIPEC drugs is unknown to patients with advanced gastric cancer, but known to doctors, investigators and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug group 1 (Experimental): hyperthermic intraperitoneal chemotherapy (HIPEC) (with paclitaxel): Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: Paclitaxel 75 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Interventions: Drug: Paclitaxel
- Drug group 2 (Experimental): hyperthermic intraperitoneal chemotherapy (HIPEC) (with lobaplatin): Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: lobaplatin 50 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Interventions: Drug: Lobaplatin
- Control group (No Intervention): hyperthermic intraperitoneal therapy (HIPET) (no drug) : Temperature Setting : 43 ± 1.0 ℃. Perfusion time: 60 min. Amount of perfusate: The perfusion fluid is based on the principle of filling the abdominal cavity and unobstructed circulation.
  Choice of perfusate: Normal saline. Drug selection and dose: no drug. Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is used as drug for hyperthermic intraperitoneal chemotherapy. Choice of perfusate: Normal saline. Drug selection and dose: Paclitaxel 75 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Arms: Drug group 1
Drug: Lobaplatin — Lobaplatin is used as drug for hyperthermic intraperitoneal chemotherapy. Choice of perfusate: Normal saline. Drug selection and dose: lobaplatin 50 mg/m2 . Treatment course: 2 times (the first time is after surgery, the second time is 48h after first time).
  Arms: Drug group 2

SUMMARY:
This study is a prospective, randomized, comparative clinical trial conducted by Wuhan Union Hospital and aim to compare the therapeutic effects of Lobaplatin and Paclitaxel in advanced gastric cancer patients with D2 surgery combined with hyperthermic intraperitoneal chemotherapy

DETAILED DESCRIPTION:
Hyperthermic intraperitoneal chemotherapy (HIPEC) is traditionally used to treat peritoneal cancer combined with cytoreductive surgery (CRS). Further, there have been lots of randomized clinical trials assessing the efficacy of surgery + HIPEC for the treatment of locally advanced gastric cancer conducted. Nonetheless, to date, the kinds, doses, combinations of HIPEC drugs are not clearly been evaluate a criterion. Thus, This study aim to compare the efficacy of Lobaplatin and Paclitaxel in advanced gastric cancer patients with D2 surgery combined with HIPEC. We plan to recruit 231 patients and divide into 3 groups, 2 drug groups and 1 control groups, radomly. all patients with advanced gastric cancer receive D2 surgery + HIPEC + SOX/XELOX chemotherapy regimen. the mainly experimental variable is HIPEC drugs and three groups employ Lobaplatin, Paclitaxel and none respectively. the endpoints of study include peritoneal metastasis, overall survival, immune status and perioperative safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. No chemoradiotherapy or other anti-tumor therapy before clinical trial performed;
2. Aged 18-75 years;
3. Male or non-pregnant or lactating women;
4. Pathological diagnosis of gastric adenocarcinoma;
5. Clinical diagnosis of T3 stage or above without distant metastasis and can be given D2 radical resection (AJCC Version 8, 2018);
6. Normal function of major organs;
7. Routine blood examinations meeting the following criteria:

   A. HB ≥ 90 g/L; B. ANC ≥ 1.5 x 10 9 /L; C. PLT ≥ 125 × 10 9 /L;
8. Chemistry indexs meeting the following criteria:

   A. TBIL < 1.5ULN; B. ALT and AST < 2.5ULN; ALB > 30 g/L C. serum Cr ≤ 1.25 ULN or endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
9. ECOG score 0-1;

Exclusion Criteria:

1. A history of other malignant tumors within 5 years;
2. Distant metastasis found during surgery;
3. Allergic to paclitaxel, lobaplatin and other related chemotherapeutic drugs;
4. Suffering from epilepsy or other mental illness, unable to control behavior;
5. Inability to tolerate surgery due to severe cardiac, pulmonary and vascular disease;
6. Pregnant or lactating women.
7. Receiving anti-cancer drug therapy from other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
peritoneal metastasis | 3-year
  peritoneal metastasis-free survival (pRFS)
overall survival | 3-year
  overall survival (OS)

SECONDARY OUTCOMES:
Number of participants with immunosuppression events as assessed by blood immunological indicators | up to 4 weeks
  Before and After Hyperthermic Intraperitoneal Chemotherapy, collect 5mL blood samples of patients for detecting immunological indicators such as CD3, CD4 and CD8 lymphocyte population; Interferon-γ; tumor necrosis factor (TNF)-α; interleukin-2, 4, 8, 10, etc
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 4 weeks
  postoperative adverse events (referring to CTCAE 5.0 [including blood routine, liver and kidney function, patient reaction to HIPEC, adverse events]) was analyzed
The positive rate of cancer cells of participants by exfoliative cytology examination | 1 week
  According to the positive rate of cancer cells measured in exfoliative cytology before and after HIPEC, the difference between the groups is analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Kaixiong Tao, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
we would like to share IPD to other researchers 1 years after clinical trial finished
Supporting Information: Study Protocol, ICF, CSR
Time Frame: we would like to share IPD to other researchers 1 years after clinical trial finished
Access Criteria: all data should not been used for commercial purpose and other private purpose and only for academic research

REFERENCES:
- [Background] Macdonald JS, Smalley SR, Benedetti J, Hundahl SA, Estes NC, Stemmermann GN, Haller DG, Ajani JA, Gunderson LL, Jessup JM, Martenson JA. Chemoradiotherapy after surgery compared with surgery alone for adenocarcinoma of the stomach or gastroesophageal junction. N Engl J Med. 2001 Sep 6;345(10):725-30. doi: 10.1056/NEJMoa010187. PMID 11547741
- [Result] Yonemura Y, de Aretxabala X, Fujimura T, Fushida S, Katayama K, Bandou E, Sugiyama K, Kawamura T, Kinoshita K, Endou Y, Sasaki T. Intraoperative chemohyperthermic peritoneal perfusion as an adjuvant to gastric cancer: final results of a randomized controlled study. Hepatogastroenterology. 2001 Nov-Dec;48(42):1776-82. PMID 11813623
- [Result] Fujimoto S, Takahashi M, Mutou T, Kobayashi K, Toyosawa T. Successful intraperitoneal hyperthermic chemoperfusion for the prevention of postoperative peritoneal recurrence in patients with advanced gastric carcinoma. Cancer. 1999 Feb 1;85(3):529-34. PMID 10091726
- [Result] Torphy RJ, Stewart C, Sharma P, Halpern AL, Oase K, Herter W, Bartsch C, Friedman C, Del Chiaro M, Schulick RD, Gleisner A, McCarter MD, Ahrendt SA. Dextrose-Containing Carrier Solution for Hyperthermic Intraperitoneal Chemotherapy: Increased Intraoperative Hyperglycemia and Postoperative Complications. Ann Surg Oncol. 2020 Dec;27(13):4874-4882. doi: 10.1245/s10434-020-08330-y. Epub 2020 Apr 19. PMID 32306237
- [Result] Hamazoe R, Maeta M, Kaibara N. Intraperitoneal thermochemotherapy for prevention of peritoneal recurrence of gastric cancer. Final results of a randomized controlled study. Cancer. 1994 Apr 15;73(8):2048-52. doi: 10.1002/1097-0142(19940415)73:83.0.co;2-q. PMID 8156509

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04808466/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/66/NCT04808466/ICF_001.pdf